CLINICAL TRIAL: NCT04367974
Title: Clinical Pharmacokinetic Study of Ceftazidime and Cefazolin in Treating CAPD-related Peritonitis
Brief Title: Clinical Pharmacokinetic Study of Ceftazidime and Cefazolin
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: WZhu
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-04

CONDITIONS: CAPD-related Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and dialysate samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: The dose of cefazolin and Ceftazidime co-administered were 20 mg /kg，they were given intraperitoneal twice daily in the first bag and the fourth bag for 5 days，and given 1g once daily in the fourth bag for 9 days. Total treatment duration was 2 weeks.
- 2: The dose of cefazolin and Ceftazidime co-administered were 20 mg /kg，and were given once daily in the fourth bag. Total treatment duration was 2 weeks.

SUMMARY:
Peritoneal dialysis-related peritonitis is a common complication of peritoneal dialysis, which is the main cause of transfer from peritoneal dialysis to hemodialysis. Guidelines for International Society for peritoneal dialysis（ISPD）published in 2016 recommend that timely and adequate use of antibiotics is the most important part of treatment. Empiric treatment should be initiated as soon as possible after obtaining microbiological specimens，then adjust the antibiotics according to culture results and drug sensitivity of bacteria. Intraperitoneal antibiotic can ensure antibiotic concentrations at the local sites of the infection are maximized，however, in patients with renal failure, the investigators should pay attention to the nephrotoxicity caused by the reduction of renal excretion，being guided by Pharmacokinetic/ Pharmacodynamic Principle on antibiotic can develop dosing recommendations to optimize antibiotic efficacy and minimize toxicity. In this study, the investigators aim to detect the concentration of ceftazidime and cefazolin in CAPD patients，so as to analyze the pharmacokinetics parameters and evaluate the rationality of the treatment.

DETAILED DESCRIPTION:
The dose of cefazolin and Ceftazidime co-administered were 20 mg /kg，they were given intraperitoneal twice daily in the first bag and the fourth bag for 5 days，and given 1g once daily in the fourth bag for 9 days. Total treatment duration was 2 weeks.

At least 1-mL serum and 5-mL dialysate samples were collected at 1, 2, 4, 6, 10, 14 days after complete instillation of the first dialysis bag containing antibiotic into the peritoneal cavity. The samples were then centrifuged at 3,000 rpm, all study samples were stored frozen (-80℃) within 1 hour after collection.

ELIGIBILITY:
Inclusion Criteria:

Maintained on continuous ambulatory PD (CAPD) for at least 1 month,all patients received 4 exchanges per day with dialysate volumes of 2 L per exchange.

1. The diagnostic criteria for CAPD-related peritonitis are as follows:

   The dialysate fluid appears cloudy and accord with the following peritonitis diagnostic criteria: (with the following two can be diagnosed) A. Clinical manifestations of peritoneics, such as abdominal pain and/or turbid flow of fluid from peritoneal dialysis; B. Perital dialysis discharge of liquid pathogen culture positive. C. The white blood cell count of perital dialysis outflow liquid were more than 0. 1 x 10 x 9/L, and the percentage of polymorphic nucleocells is more than 50% (peritoneal dialysis fluid remains in the abdominal cavity for at least 2 hours for more than 2 hours);
2. No urine (less than 100ml per 24h).
3. Age range form 15 years old to 70 years old, gender is not limited;
4. Understand and agree to this clinical trial study.

Exclusion Criteria:

1. With a clear history of cephalosporine drug allergy or hypersensitivity;
2. Received antibiotic treatment within 1 week prior to entering the study;
3. Pregnant and lactating women;
4. Sepsis;
5. Patients with celiac malignancy;
6. The patient is unable to cooperate or unwilling to accept the test.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CAPD-related peritonitis patients who accord with the inclusion Criteria and without the exclusion Criteria.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
concentration of ceftazidime and cefazolin | 2 weeks
  Cefazolin and ceftazidime were measured by LC-MS. The lower limit of quantitation for cefazolin and ceftazidime was 0.05 -1.0 μg /ml.

CONTACTS AND LOCATIONS:
Locations (1):
- the fifth affiliated hospital of SUN YAT-SEN university, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li PK, Szeto CC, Piraino B, de Arteaga J, Fan S, Figueiredo AE, Fish DN, Goffin E, Kim YL, Salzer W, Struijk DG, Teitelbaum I, Johnson DW. ISPD Peritonitis Recommendations: 2016 Update on Prevention and Treatment. Perit Dial Int. 2016 Sep 10;36(5):481-508. doi: 10.3747/pdi.2016.00078. Epub 2016 Jun 9. No abstract available. PMID 27282851
- [Result] Htay H, Cho Y, Pascoe EM, Hawley C, Clayton PA, Borlace M, Badve SV, Sud K, Boudville N, McDonald SP, Johnson DW. Outcomes of Acinetobacter Peritonitis in Peritoneal Dialysis Patients: A Multicenter Registry Analysis. Perit Dial Int. 2018 Jul-Aug;38(4):257-265. doi: 10.3747/pdi.2017.00199. Epub 2018 Feb 7. PMID 29437143
- [Result] Ranganathan D, Varghese JM, Fassett RG, Lipman J, D'Intini V, Healy H, Roberts JA. Optimising intraperitoneal gentamicin dosing in peritoneal dialysis patients with peritonitis (GIPD) study. BMC Nephrol. 2009 Dec 16;10:42. doi: 10.1186/1471-2369-10-42. PMID 20003546
- [Result] Manley HJ, Bailie GR. Treatment of peritonitis in APD: pharmacokinetic principles. Semin Dial. 2002 Nov-Dec;15(6):418-21. doi: 10.1046/j.1525-139x.2002.00103.x. PMID 12437537
- [Result] McKinnon PS, Paladino JA, Schentag JJ. Evaluation of area under the inhibitory curve (AUIC) and time above the minimum inhibitory concentration (T>MIC) as predictors of outcome for cefepime and ceftazidime in serious bacterial infections. Int J Antimicrob Agents. 2008 Apr;31(4):345-51. doi: 10.1016/j.ijantimicag.2007.12.009. Epub 2008 Mar 4. PMID 18313273
- [Result] Cardone KE, Grabe DW, Zasowski EJ, Lodise TP. Reevaluation of ceftazidime dosing recommendations in patients on continuous ambulatory peritoneal dialysis. Antimicrob Agents Chemother. 2014;58(1):19-26. doi: 10.1128/AAC.00873-13. Epub 2013 Oct 14. PMID 24126585
- [Result] Tosukhowong T, Eiam-Ong S, Thamutok K, Wittayalertpanya S, Na Ayudhya DP. Pharmacokinetics of intraperitoneal cefazolin and gentamicin in empiric therapy of peritonitis in continuous ambulatory peritoneal dialysis patients. Perit Dial Int. 2001 Nov-Dec;21(6):587-94. PMID 11783768
- [Result] Booranalertpaisarn V, Eiam-Ong S, Wittayalertpanya S, Kanjanabutr T, Na Ayudhya DP. Pharmacokinetics of ceftazidime in CAPD-related peritonitis. Perit Dial Int. 2003 Nov-Dec;23(6):574-9. PMID 14703199
- [Result] Grabe DW, Bailie GR, Eisele G, Frye RF. Pharmacokinetics of intermittent intraperitoneal ceftazidime. Am J Kidney Dis. 1999 Jan;33(1):111-7. doi: 10.1016/s0272-6386(99)70265-9. PMID 9915275